CLINICAL TRIAL: NCT02542761
Title: Comparative Performance of Dynamic Elastic Response Feet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kenton R. Kaufman, Ph.D., PI, Mayo Clinic
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15-001367
Record Dates: First submitted 2015-06-15; First posted 2015-09-07 (Estimated); Results first posted 2017-09-08 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Transtibial Amputation - Unilateral

STUDY DESIGN:
Intervention Model Description: This was a repeated measures cross-over trial whereby only the prosthetic foot was changed. Each subject was tested using their current carbon-fiber prosthetic foot (CFPF), and the fiberglass prosthetic foot (FPF). Half of the subjects began the study on the CFPF while the other half began on the FPF. Each subject was given an acclimation period of 4 weeks before testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CFPF first, then FPF (Experimental): After a 4 week acclimation period, subjects were studied on their current carbon fiber composite foot (CFPF), followed by another 4 week acclimation period, then studied on the study provided fiberglass composite foot (FPF).
  Interventions: Device: Fiberglass Composite foot; Device: Carbon Fiber Composite Foot
- FPF first, then CFPF (Experimental): After a 4 week acclimation period, subjects were studied on the study provided fiberglass composite foot (FPF), followed by another 4 week acclimation period, then studied on their current carbon fiber composite foot (CFPF).
  Interventions: Device: Fiberglass Composite foot; Device: Carbon Fiber Composite Foot

INTERVENTIONS:
Device: Fiberglass Composite foot — The Rush foot is a fiberglass composite energy storage and return prosthetic foot.
  Other Names: Rush Foot
Device: Carbon Fiber Composite Foot — All types of currently commercially available carbon fiber energy storage and return prosthetic feet will be considered appropriate.
  Other Names: Otto Bock Triton; Ossur Variflex; Ossur Variflex EVO; Ossur Reflex Shock; Freedom Renegade; Freedom Pacifica; Freedom Thrive with Vertical Shock; Freedom Highlander; Freedom Agilix

SUMMARY:
The purpose of this study was to compare the functional performance of individuals with transtibial amputation using two types of prosthetic foot designs: carbon fiber vs. fiberglass composite.

DETAILED DESCRIPTION:
Recently, a new type of prosthetic foot has appeared on the market. This device is composed of a fiberglass composite material. Knowledge is lacking regarding the performance characteristics of this new device. Comprehensive studies are needed to form a solid basis for prosthetic prescription. The current study sought to understand the experience of community-living, transtibial amputees using this prosthetic foot. Specifically, the biomechanical performance of this device were compared to existing conventional dynamic elastic response (DER) technology in a controlled laboratory setting. The investigators hypothesized that the fiberglass composite material provided more energy return and improved ankle kinematics performance.

The study design was a repeated measures cross-over trial whereby only the prosthetic foot was changed. Each subject was tested using their current carbon-fiber energy storage and return prosthetic foot (CFPF) and the fiberglass composite energy storage and return prosthetic foot (Rush, Ability Dynamics) (FPF). Half of the subjects began the study on the CFPF while the other half began on the FPF. All types of CFPF were used in this study. Each subject was given an acclimation period (about 4 weeks) before testing, which was consistent with other similar studies. The same socket and suspension were used throughout the study in order to eliminate these confounding variables.

A 10 camera, high resolution motion capture system with a set of 51 reflective markers was used to capture whole-body motion. Three-dimensional marker trajectory data was collected at 120 Hz and filtered using a fourth-order Butterworth low-pass filter with a cutoff frequency of 8 Hz. The standard Helen Hayes marker set and some additional markers were applied to the subject. Additional markers included an anterior pylon marker, medial pylon marker, lateral pylon marker, right and left medial calcaneus markers, and right and left lateral calcaneus markers. In addition, left and right medial knee markers were used for establishing the knee joint centers and were then removed for the walking trails. Subjects wore standard laboratory athletic shoes for all walking trials. All of the markers associated with the foot were placed on the outside of the subject's shoes.

Following the application of the reflective marker set, the subject performed tests while walking over level ground at a self-selected and normalized speed as well as up and down a 10 degree inclined ramp. The normalized speed controlled for leg length by normalizing to a Froude (Fr) number of 0.25 where Fr = v^2/gl, and v is the walking speed, g is the gravitational constant, and l is the leg length using the greater trochanter height as leg length. Timing gates were used to control the walking speed. Simultaneously, ground reaction force data was collected from force plates at a sampling rate of 600 Hz. Data from these force plates was time-synchronized with the motion cameras. The ramp had a force plate embedded within the ramp.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputee
* Currently using a carbon fiber prosthetic (DER) foot for at least the last 6 months
* Stable stump volume over the past 6 months
* Medicare Functional Classification Level K3 or K4

Exclusion Criteria:

* Neuromuscular problems such as previous stroke or contralateral amputation
* Use of gait aids for ambulation
* Undergoing dialysis
* Poor prosthetic socket fit or stump problems (e.g., skin breakdown)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenton R Kaufman, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kaufman KR, Bernhardt K. Functional performance differences between carbon fiber and fiberglass prosthetic feet. Prosthet Orthot Int. 2021 Jun 1;45(3):205-213. doi: 10.1097/PXR.0000000000000004. PMID 33856155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at Mayo Clinic in Rochester, Minnesota.
Period: Acclimation Period 1
Arm/Group | CFPF First, Then FPF | FPF First, Then CFPF
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: First Intervention
Arm/Group | CFPF First, Then FPF | FPF First, Then CFPF
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Acclimation Period 2
Arm/Group | CFPF First, Then FPF | FPF First, Then CFPF
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | CFPF First, Then FPF | FPF First, Then CFPF
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups studying CFPF first and FPF first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29 (7)

OUTCOME MEASURES:

1. Primary Outcome: Peak Ankle Dorsiflexion During Stance
Description: The peak ankle dorsiflexion is the peak ankle backward flexion or bending when walking.
Time Frame: After approximate 4 week acclimation period
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Carbon Fiber Prosthetic Foot (CFPF): All types of currently commercially available carbon fiber energy storage and return prosthetic feet will be considered appropriate.
- Fiberglass Prosthetic Foot (FPF): The Rush87 foot is a fiberglass composite energy storage and return prosthetic foot.
Arm/Group | Carbon Fiber Prosthetic Foot (CFPF) | Fiberglass Prosthetic Foot (FPF)
Number analyzed (Participants) | 10 | 10
degrees
  Level ground, controlled speed | 18.871 (2.549) | 22.023 (2.654)
  Level ground, self-selected speed | 18.657 (2.818) | 22.016 (2.638)
  Ramp Down | 17.09 (3.22) | 19.98 (3.18)
  Ramp Up | 20.45 (4.38) | 23.80 (4.09)

2. Secondary Outcome: Peak Ankle Plantar Flexor Moment During Stance
Description: Peak ankle plantar flexor moment means the peak force of the movement of the foot in which the foot or toes flex downward toward the sole. The unit of measurement for this variable is Nm/kg = 1 nanometer / (kilogram unit).
Time Frame: After approximate 4 week acclimation period
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | Carbon Fiber Prosthetic Foot (CFPF) | Fiberglass Prosthetic Foot (FPF)
Number analyzed (Participants) | 10 | 10
Nm/kg
  Level ground, self selected speed | 1.3446 (0.1306) | 1.4451 (0.2333)
  Level ground, normalized speed | 1.3732 (0.1915) | 1.4418 (0.2361)
  Ramp Down | 1.0989 (0.1765) | 1.1662 (0.2197)
  Ramp Up | 1.4787 (0.2244) | 1.5251 (0.2922)

3. Secondary Outcome: Peak Ankle Power Generation
Description: Joint power (P) is the "dot product" of the moment (M) at the joint and the angular velocity (w) of the distal segment with respect to the proximal segment (i.e., P = M · w). Depending on the direction of the moment and the direction of the angular velocity, the power can be positive or negative. If the signs for the moment and angular velocity are both positive or both negative, the power is positive. If the signs for the moment and angular velocity are different, the power is negative. The unit of measurement for this variable is W/kg = watts/kilogram.
Time Frame: After approximate 4 week acclimation period
Measure: Mean (Standard Deviation); unit: W/kg
Arm/Group | Carbon Fiber Prosthetic Foot (CFPF) | Fiberglass Prosthetic Foot (FPF)
Number analyzed (Participants) | 10 | 10
W/kg
  Level ground, controlled speed | 1.130 (0.321) | 1.605 (0.371)
  Level ground, self-selected speed | 1.080 (0.318) | 1.475 (0.347)
  Ramp Down | 0.979 (0.347) | 1.292 (0.323)
  Ramp Up | 0.999 (0.416) | 1.331 (0.491)

4. Secondary Outcome: Peak Knee Flexion During Swing
Description: A gait cycle is the period of time for one stride, that is, the time from one event (usually initial foot contact) to the next occurrence of the same event with the same foot. For each leg, the gait cycle can be divided into a stance phase and a swing phase. This variable is measuring the angle of knee flexion during the swing phase.
Time Frame: After approximate 4 week acclimation period
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Carbon Fiber Prosthetic Foot (CFPF) | Fiberglass Prosthetic Foot (FPF)
Number analyzed (Participants) | 10 | 10
degrees
  Level ground, controlled speed | 69.61 (4.92) | 71.52 (7.70)
  Level ground, self-selected speed | 67.38 (4.72) | 70.08 (6.73)
  Ramp Down | 72.42 (5.75) | 73.57 (6.44)
  Ramp Up | 69.63 (6.91) | 71.45 (7.37)

5. Secondary Outcome: Time of Peak Knee Flexion During Swing
Description: A gait cycle is the period of time for one stride, that is, the time from one event (usually initial foot contact) to the next occurrence of the same event with the same foot. For each leg, the gait cycle can be divided into a stance phase and a swing phase. This variable is expressed as a percentage of the gait cycle.
Time Frame: After approximate 4 week acclimation period
Measure: Mean (Standard Deviation); unit: percentage of gait cycle
Arm/Group | Carbon Fiber Prosthetic Foot (CFPF) | Fiberglass Prosthetic Foot (FPF)
Number analyzed (Participants) | 10 | 10
percentage of gait cycle
  Level ground, controlled speed | 71.841 (1.782) | 72.077 (2.018)
  Level ground, self-selected speed | 72.132 (1.975) | 72.293 (2.087)
  Ramp Down | 67.794 (2.409) | 67.194 (1.773)
  Ramp Up | 75.883 (2.871) | 75.653 (2.481)

6. Secondary Outcome: Patient Satisfaction as Measured by the Prosthesis Evaluation Questionnaire (PEQ)
Description: The PEQ is a self-administered questionnaire composed of nine scales computed from forty-two items (ambulation, appearance, frustration, perceived response, residual limb health, social burden, sounds, utility, well being). Each question uses a visual analog scale format, scored as a continuous numerical variable measured as the distance in millimeters from the left endpoint of the measured from the left (0-100). The 0 side of the scale is very negative (terrible) and the 100 side of the scale is very positive (excellent). Each scale is reported separately, with a higher score indicating more satisfaction with the prosthesis itself or quality of life.
Time Frame: After approximate 4 week acclimation period
Population: Some participants did not complete some of the scales in the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Prosthetic Foot (CFPF) | Fiberglass Prosthetic Foot (FPF)
Number analyzed (Participants) | 10 | 10
units on a scale
  Ambulation | 79.64 (16.49) | 84.74 (14.01)
  Appearance | 77.89 (17.51) | 85.83 (13.80)
  Frustration | 78.25 (14.94) | 83.00 (22.66)
  Perceived Response: number analyzed (Participants) | 9 | 9
  Perceived Response | 95.71 (7.18) | 93.71 (7.62)
  Residual Limb Health | 75.78 (14.99) | 77.10 (9.21)
  Social Burden: number analyzed (Participants) | 10 | 9
  Social Burden | 91.18 (14.48) | 92.57 (14.59)
  Sounds | 66.45 (27.24) | 74.50 (24.57)
  Utility | 73.31 (20.93) | 83.97 (14.36)
  Well Being | 84.15 (15.39) | 92.85 (8.95)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Carbon Fiber Prosthetic Foot (CFPF) | Fiberglass Prosthetic Foot (FPF)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes